CLINICAL TRIAL: NCT07016516
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single and Multiple Doses Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PRT-064040 Nasal Spray in Healthy Adult Subjects
Brief Title: A Study to Learn About PRT-064040 Nasal Spray in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Purity Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-PRT-064-101
Record Dates: First submitted 2025-05-27; First posted 2025-06-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single dose of PRT-064040 nasal spray (Experimental)
  Interventions: Drug: PRT-064040 nasal spray
- Single dose of Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Multiple doses of PRT-064040 nasal spray (Experimental)
  Interventions: Drug: PRT-064040 nasal spray
- Multiple doses of Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRT-064040 nasal spray — A single dose of PRT-064040 nasal spray at one of six dose levels
  Arms: Single dose of PRT-064040 nasal spray
Drug: Placebo — A single dose of Placebo at one of six dose levels
  Arms: Single dose of Placebo
Drug: PRT-064040 nasal spray — Multiple doses of PRT-064040 nasal spray at one of two dose levels, administered once daily (QD) for a total of 7 consecutive days
  Arms: Multiple doses of PRT-064040 nasal spray
Drug: Placebo — Multiple doses of Placebo at one of two dose levels, administered once daily (QD) for a total of 7 consecutive days
  Arms: Multiple doses of Placebo

SUMMARY:
This trial is a Phase I, single-center, randomized, double-blind, placebo-controlled study conducted in healthy Chinese adult subjects.

The purpose of this study is to learn about:

* Safety and tolerability of PRT-064040 nasal spray in healthy adult subjects.
* Pharmacokinetics after single and multiple dose of PRT-064040 nasal spray in healthy Chinese adult subjects.

This study is divided into two parts:

* Eligible subjects in Part A will receive a single dose of PRT-064040 nasal spray or placebo.
* Eligible subjects in Part B will receive multiple doses of PRT-064040 nasal spray or placebo, administered once daily (QD) for a total of 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female Chinese adults aged ≥18 years and ≤55 years.
2. Body Mass Index of 18 to 28 kg/m^2; and a total body weight ≥50 kg for males and ≥45 kg for females.

Exclusion Criteria:

1. History of allergy to any medications, foods, or other substances.
2. History or presence of any severe diseases that are considered clinically significant by the investigator.
3. Any clinically significant abnormal laboratory test results or positive test.
4. Any nasal conditions or diseases that, in the investigator's judgment, may significantly affect the administration or absorption of a nasal product.
5. Standard 12-Lead Electrocardiogram that demonstrates clinically relevant abnormalities.
6. Pregnant or breastfeeding women, or those with a positive pregnancy test result during screening.
7. Positive urine drug screen, alcohol breath test, or nicotine test.
8. History of significant alcohol abuse or drug abuse.
9. Donation or loss of blood of approximately 400 mL or more within 3 months prior to dosing.
10. Previous participation in another clinical trial and receiving the investigational drug within 3 months prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-06-07 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | From first dose to maximum of 2 days post last dose administration

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: Cmax | Up to 2 days post last dose administration
Pharmacokinetic Parameters: Tmax | Up to 2 days post last dose administration
Pharmacokinetic Parameters: AUC | Up to 2 days post last dose administration
Pharmacokinetic Parameters: Half life | Up to 2 days post last dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No